CLINICAL TRIAL: NCT03326518
Title: An Open, Randomized, Controlled, Single Centre Trial to Evaluate CT Image Quality and Diagnostic Feasibility of Lumentin® 44, in Comparison With Omnipaque and Movprep.
Brief Title: A Randomized, Controlled Trial to Evaluate CT Image Quality Lumentin® 44
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary objective reached
Sponsor: Lument AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LUM-001
Record Dates: First submitted 2017-10-17; First posted 2017-10-31 (Actual); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-05

CONDITIONS: Subjects Referred to CT-examination of the Abdomen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumentin® 44 (Experimental): Contrast agent
  Interventions: Diagnostic Test: Lumentin® 44
- Diluted Omnipaque® (Active Comparator): Contrast agent
  Interventions: Diagnostic Test: Diluted Omnipaque®
- Movprep® (Active Comparator): Contrast agent
  Interventions: Diagnostic Test: Movprep®

INTERVENTIONS:
Diagnostic Test: Lumentin® 44 — Contrast agent
  Arms: Lumentin® 44
Diagnostic Test: Diluted Omnipaque® — Contrast agent
  Arms: Diluted Omnipaque®
Diagnostic Test: Movprep® — Contrast agent
  Arms: Movprep®

SUMMARY:
Subjects referred for abdominal or thoracoabdominal CT-examination will be randomised to either the three contrast agents Lumentin® 44, Omnipaque® or Movprep. The difference in contrast density, as observed in the CT-examination, between lumen and wall (mucosal lining) will be compared by the three contrast agents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender at least 18 years at the time of signing the informed consent.
* Having a clinical indication for CT-examination of the abdomen

Exclusion Criteria:

* IV administration of iodine is contraindicated
* Known allergy to egg albumen
* Clinical suspicion, according to medical record, of fistula formation and/or leakage
* Referral indication of small bowel disease(s)
* Having known manifest thyrotoxicosis
* Having known phenylketonuria
* Having known Glucose-6-phosphatase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leander, Ass. Prof., Principal Investigator — Skanes University Hospital
Locations (1):
- Department of medical imaging and function, Malmo, Sweden

REFERENCES:
- [Derived] Leander P, Stathis G, Casal-Dujat L, Boman K, Adnerhill I, Marsal J, Book O, Fork T. A novel food-based negative oral contrast agent compared with two conventional oral contrast agents in abdominal CT: a three-arm parallel blinded randomised controlled single-centre trial. Eur Radiol Exp. 2022 Apr 5;6(1):15. doi: 10.1186/s41747-022-00267-z. PMID 35378633

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Started | 19 | 12 | 14
Completed | 16 | 12 | 13
Not Completed | 3 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep® | Total
Number analyzed (Participants) | 19 | 12 | 14 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 8 | 19
  >=65 years | 13 | 7 | 6 | 26
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 6 | 5 | 8 | 19
  65-84 years | 13 | 6 | 6 | 25
  85 years and over | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 8 | 27
  Male | 8 | 4 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 19 | 12 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Relative Mean Difference in Contrast Density
Description: difference in contrast density between lumen and wall (mucosal lining)
Time Frame: Day 1
Population: Two patients in the Lumentin group withdrew prior to contrast agent intake and were withdrawn from the efficacy analysis.
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Hounsfield units | 484.0 (192.4) | 122.1 (81.4) | 64.5 (15.9)

2. Secondary Outcome: Bowel Filling Properties, Extension
Description: The bowel filling agent was distributed along the length of small bowel, i.e. the extension. The filling of each of the 5 selected sub-segments of the small bowel in terms of extension was examined on the CT-scan by 2 investigators, independently of each other, and graded using Likert scales between 1 and 9.
  Extension scale:
  1. No sign of contrast agent
  2. Trace of contrast agent filling
  3. Segment filled to ca. 25%
  4. Segment filled to >25% but <50%
  5. Filled to segment filled to 50%
  6. Segment filled > 50% but <75%
  7. Segment filled to ca. 75%
  8. Segment filled to >75% but <100%
  9. Segment filled to 100% The evaluation was made by 2 independent radiology experts. The Extension score is the sum of the grades in each sub-segment from both evaluations and hence range from 10 to 90.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Likert Scale score
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Likert Scale score | 63.0 (21.7) | 61.2 (15.9) | 71.8 (10.6)

3. Secondary Outcome: Bowel Filling Properties, Distension
Description: The bowel filling agent caused a local widening of the bowel loop, distension. The filling of each of the 5 selected sub-segments of the small bowel in terms of distension was examined on the CT-scan by both the 2 investigators independently of each other, and graded using Likert scales between 1 and 9.
  Distension scale:
  1. No identifiable contrast agent
  2. A minimal amount of contrast agent is identified
  3. Small amount of contrast agent, insufficient for placing a ROI of 6 mm
  4. Amount of contrast agent just allowing for a ROI of 6 mm
  5. Medium filled bowel loop
  6. Slightly better than grade 5
  7. Good filling
  8. Optimal filling
  9. Excellent or almost over distended The evaluation was made by 2 independent radiology experts. The Distension score is the sum of the grades in each sub-segment from both evaluations and hence range from 10 to 90.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Likert Scale score
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Likert Scale score | 48.1 (18.1) | 47.0 (12.2) | 54.7 (8.6)

4. Secondary Outcome: Diagnostic Ability When Examining Abdominal CT
Description: Diagnostic ability when examining Abd-CT was assessed on the CT-scan by the 2 investigators independently of each other.
  The following features were assessed:
  * Small bowel appearance
  * Parenchymal organs, i.e. Pancreas, ovaries, urinary bladder
  * Mesenterium and omentum using a Likert scales of 1-9 ranging, where:
    1.Impossible to observe details
    5. Medium
    9. Excellent resolution
  The evaluation was made by 2 independent radiology experts. The Diagnostic ability score is the sum of the scores of each feature from both evaluations and hence range from 6 to 54.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Likert Scale score
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Likert Scale score | 43.1 (4.8) | 39.9 (5.9) | 41.4 (4.4)

5. Secondary Outcome: Degradation of Contrast Agent (Lumentin® 44)
Description: Degradation of Lumentin 44 was founded on the 2 characteristics; coalescence and syneresis or drainage.
  Coalescence:
  0. No bubbles visually detectable at the CT-scan
  1. Bubbles visually detectable at the CT-scan
  Syneresis or drainage:
  0. No syneresis or drainage, i.e. separation of air and liquid phases, observed
  1. Syneresis or drainage observed Signs of degradation were assessed on the CT-scan, by both Investigator and Sub-Investigator, independently of each other, in each of the 5 selected sub-segments of the small bowel.
  The degradation of contrast agents score is the sum of the scores in each sub-segment and range from 0 to 10.
Time Frame: Day 1
Population: Lumentin 44 is a foam containing air, and it could be suspected that the air bubbles would not withstand the condition in the stomach/intestines. Therefore, the end point Degradation of Contrast Agent was only valid for Lumentin 44 and it was included to prove the resisting power of Lumentin 44 and not to compare the IMP with Omnipaque or Movprep.
Measure: Mean (Standard Deviation); unit: Scores on a scale (0-10)
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 0 | 0
Scores on a scale (0-10) | 0.647 (0.996) |  |

6. Secondary Outcome: Subjects' Assessment of Taste of the Contrast Agent
Description: The subjects assessed taste on a five degree-scale:
  1. Very negative
  2. Negative
  3. Neutral
  4. Positive
  5. Very positive
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Score (1-5)
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Score (1-5) | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 5.0] | 2.5 [1.0 to 4.0]

7. Secondary Outcome: Subjects' Assessment of Smell of the Contrast Agent
Description: as for outcome 6
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Score (1-5)
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Score (1-5) | 4.0 [3.0 to 5.0] | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 5.0]

8. Secondary Outcome: Subjects' Assessment of Consistency of the Contrast Agent
Description: as for outcome 6
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Score (1-5
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Score (1-5 | 3.0 [2.0 to 4.0] | 4.0 [3.0 to 5.0] | 3.0 [2.0 to 4.0]

9. Secondary Outcome: Subjects' Assessment of Ability to Swallow the Contrast Agent
Description: as for outcome 6
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Score (1-5)
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Score (1-5) | 3.0 [2.0 to 4.0] | 5.0 [2.0 to 5.0] | 3.0 [1.0 to 5.0]

10. Secondary Outcome: Subjects' Assessment of Fullness After Drinking the Contrast Agent
Description: as for outcome 6
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Score (1-5)
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
Number analyzed (Participants) | 17 | 12 | 14
Score (1-5) | 2.0 [1.0 to 4.0] | 3.0 [2.0 to 4.0] | 3.0 [1.0 to 5.0]

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Lumentin® 44 | Diluted Omnipaque® | Movprep®
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 7/18 | 7/12 | 8/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumentin® 44 (N=18) | Diluted Omnipaque® (N=12) | Movprep® (N=14)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 6 (6)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT03326518/Prot_SAP_000.pdf